CLINICAL TRIAL: NCT01687673
Title: Phase II Trial of the Combination of Temsirolimus and Sorafenib in Advanced Hepatocellular Carcinoma
Brief Title: Phase II Combination of Temsirolimus and Sorafenib in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Robert H. Lurie Cancer Center (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 124511; NCI-2012-02021 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Results first posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Advanced HCC; Temsirolimus; TORISEL; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — temsirolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Combination temsirolimus plus sorafenib
  Interventions: Drug: Temsirolimus; Drug: Sorafenib:

INTERVENTIONS:
Drug: Temsirolimus — 10 mg weekly will be administered intravenously over 30 to 60 minutes using an infusion pump starting on Cycle 1, Day 1 of study enrollment.
Drug: Sorafenib: — 200 mg tablet twice daily starting on Cycle 1, Day 1 of study enrollment after completion of temsirolimus infusion.

SUMMARY:
This Phase II trial is being developed following the completion of a Phase I study of the combination of temsirolimus and sorafenib in 25 first-line therapy patients with advanced hepatocellular carcinoma (December 2009 through April 2012). The maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of the combination of temsirolimus is 10 mg IV weekly plus sorafenib 200 mg (oral, twice daily).

DETAILED DESCRIPTION:
The hypothesis of this single-arm phase II study is that the combination of temsirolimus and sorafenib will achieve a clinically-meaningful median time to progression (TTP) of at least 6 months, with null hypothesis of less than or equal to 3 months, in first-line systemic therapy for patients with advanced Hepatocellular carcinoma (HCC). A randomized trial would be required to formally compare the efficacy of this combination to sorafenib alone and will be indicated if this phase II study achieves a median TTP of at least 6 months. An interim safety analysis will employ stopping rules after 30% of planned patients have been treated with at least one dose of protocol therapy to ensure the combination does not confer excessive toxicity.

A key aspect of this study will be the requirement of histologic confirmation along with adequate archival tissue for correlative tissue analyses to explore new biomarkers of response to mammalian target of rapamycin (mTOR) inhibition. Circulating biomarker data including enumeration of circulating tumor cells (CTC) and measurement of the tumor marker Alpha-fetoprotein (AFP) will be performed at specific time points to evaluate for predictive value. Specimen banking of tissue, serum, and peripheral blood mononuclear cells will be undertaken to enable future novel biomarker studies. Modified RECIST will be performed in addition to standard RECIST 1.1 to explore for improved imaging predictors of response.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients must have histologically diagnosed American Joint Committee on Cancer (AJCC) stage II, III, or IV hepatocellular carcinoma (HCC) not eligible for curative resection, transplantation, or ablative therapies
2. Radiographically measurable disease by RECIST version 1.1 in at least one site not previously treated with chemoembolization, radioembolization, or other local ablative procedures (i.e. must have at least one measurable target lesion, either within the liver or in a measurable metastatic site); a new area of tumor progression within or adjacent to a previously-treated lesion, if clearly measurable by a Radiologist, is acceptable
3. No prior systemic cytotoxic chemotherapy or targeted therapy (including sorafenib) for HCC
4. Prior chemoembolization, local ablative therapies, or hepatic resection permitted if completed ≥ 4 weeks prior to study enrollment if patient has recovered with ≤ grade 1 toxicity and if measurable disease (criterion 2) is present
5. Prior radiation for bone or brain metastases is permitted if patient is now asymptomatic and has completed all radiation and steroid therapy (if applicable) for brain or bone metastases ≥ 2 weeks prior to study enrollment.
6. Age ≥ 18 years.
7. Child-Pugh score of A or B with ≤ 7 points and meeting laboratory eligibility for all parameters
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Life expectancy greater than 3 months
10. Treatment with appropriate antiviral therapy for patients with active hepatitis B Virus (HBV) infection is required
11. Treatment for clinically-significant hyperglycemia, hyperlipidemia, or hypertension that develops on study is required
12. Baseline blood pressure must be adequately controlled with or without antihypertensive medications prior to enrollment (systolic ≤ 150 mm Hg, diastolic ≤ 90 mm Hg)
13. Baseline cholesterol must be < 350 mg/dL and triglycerides < 300 mg/dL (with or without the use of antihyperlipidemic medications)
14. Baseline fasting blood glucose must be ≤ 140 mg/dL and hemoglobin A1c less than 7.5% (with or without the use of anti-diabetic medications)
15. Adequate baseline organ and marrow function as defined below

    Adequate bone marrow function:

    absolute neutrophil count > = 1,000/microliter (mcL) platelets ≥ 75,000/mcL hemoglobin ≥ 8.5 g/dL

    Adequate hepatic function:

    total bilirubin ≤ 2 mg/dL or ≤ 1.5 times ULN aspartate aminotransferase (AST) / serum glutamic-oxaloacetic transaminase (SGOT) & alanine aminotransferase (ALT) / serum glutamic-pyruvic transaminase (SGPT) ≤ 5 X upper limit of normal (ULN) International Normalized Ratio (INR) <=1. 5 X ULN

    Adequate renal function:

    albumin ≥ 2.8 g/dL creatinine ≤1. 5 X ULN
16. Able to tolerate oral therapy.
17. Ability to understand and willingness to provide informed consent, and the willingness to comply with the requirements of the protocol. Informed consent may be obtained with the assistance of a medical translator according to institutional policies.
18. The effects of temsirolimus on the developing human fetus are unknown. For this reason and because sorafenib - also being used in this trial - is known to be teratogenic, women of child-bearing potential must have a negative pregnancy test within 14 days of study enrollment.

    Also, women of child-bearing potential and men must agree to use two methods adequate contraception (hormonal plus barrier or two forms of barrier) or abstinence prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she needs to inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, or be surgically sterile, for the duration of study participation, and for 3 months after completion of study drug administration.
19. Eligibility of patients receiving any medications or substances known to affect or with potential to affect the activity or pharmacokinetics of temsirolimus and/or sorafenib will be determined following review of the case by the Study Chair. Efforts should be made to switch patients who are taking enzyme-inducing anti-convulsant agents to other medications.
20. mixed histology (mixed HCC-cholangiocarcinoma) tumors if deemed appropriate for HCC therapy by treating MD

EXCLUSION CRITERIA:

1. Mixed tumor histology or fibrolamellar variant tumors are excluded.
2. Prior systemic or antiangiogenic therapy for HCC (including thalidomide, sorafenib, sunitinib, or bevacizumab). Prior systemic therapy for other diagnoses is permitted if greater than 6 months have elapsed since last dose, any prior toxicity has recovered to ≤ grade 1 by CTCAE v4.0, and treatment was not discontinued for toxicity.
3. Prior treatment with mTOR inhibitor or other molecularly targeted therapy.
4. Prior systemic cytotoxic therapies for HCC (chemoembolization is permitted if inclusion criteria are met).
5. Treatment with other investigational agents.
6. Immunosuppressive medications including systemic corticosteroids unless used for adrenal replacement, appetite stimulation, acute therapy for asthma or bronchitis exacerbation (≤ 2 weeks), or antiemesis
7. Patients with known HIV infection are ineligible due to risk of pharmacokinetic interactions between anti-retroviral therapy and the study drugs, as well as potential for significant immunosuppression and serious infections with mTOR inhibition.
8. Patients who have undergone liver transplantation are excluded.
9. Uncontrolled hypertension (> 150/90 mmHg).
10. Uncontrolled hyperlipidemia (total cholesterol > 350 or triglycerides > 300).
11. Symptomatic brain or bone metastases; prior radiation and/or steroid therapy for brain or bone metastases (if applicable) must be completed ≥ 2 weeks prior to study enrollment.
12. History of seizure disorder requiring antiepileptic medication or brain metastases with seizures.
13. Serious non-healing wound, ulcer, bone fracture, or abscess.
14. Major surgical procedure less than 4 weeks from start of protocol treatment.
15. Patients requiring chronic anticoagulation with warfarin are excluded. Patients treated with low molecular weight heparin or unfractionated heparin are eligible if on a stable dose without evidence of clinically significant bleeding for at least 2 weeks prior to enrollment.
16. Active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ. (Patients with history of malignancy are not considered to have a "currently active" malignancy if they have completed therapy and are now considered by their physician to be at less than 30% risk for relapse.)
17. Uncontrolled intercurrent illness including, but not limited to: Ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled peripheral vascular disease, myocardial infarction within preceding 12 months, cerebrovascular accident within preceding 12 months, pulmonary disease impairing functional status or requiring oxygen, impairment in gastrointestinal function that may affect or alter absorption of oral medications (such as malabsorption or history of gastrectomy or bowel resection).
18. Patients will be excluded if there is any history of allergic reaction(s) attributed to compounds of similar composition to temsirolimus, sorafenib, their metabolites, or any component of their formulation (including excipients and polysorbate 80). This includes hypersensitivity to macrolide antibiotics due to potential for cross-reactivity with temsirolimus.
19. Pregnant or lactating women are excluded from this study because temsirolimus and sorafenib are drugs with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with temsirolimus or sorafenib, breastfeeding should be discontinued if the mother is receiving temsirolimus/sorafenib treatment.
20. Patients who require prohibited medications with potential for serious interactions with protocol therapy, and who cannot have therapeutic substitution are excluded. Patients receiving any medications or substances that are inhibitors or inducers of CYP450 enzyme(s) are ineligible. Lists of prohibited medications and substances known, or with the potential to interact with the specified CYP450 enzyme(s) isoenzymes are provided in Appendices 6-9 Prohibited Medications
21. Psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10-05 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Kelley, MD, Study Chair — University of California, San Francisco; Kate Kelley, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 29
Completed (One patient was removed for hepatic decompensation before starting study treatment) | 28
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 61 [33 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Baseline Alpha-fetoprotein (AFP) [Count of Participants; unit: Participants]
  < 400 nanograms per millilitre (ng/mL) | 20
  >= 400 ng/mL | 9

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression (TTP)
Description: Median TTP will be calculated in months from date of first dose of protocol therapy to date of removal from study for progression, where progression is defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as at least a 20% increase in the sum of the longest diameter of the target lesions (SLD), taking as reference the smallest sum of the SLD recorded since the treatment started and minimum 5 millimeter (mm) increase over the nadir, or the appearance of one or more new lesions for target lesions and/or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions . Kaplan-Meier methods will be used to summarize the primary endpoint
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 28
months | 3.7 [2.2 to 5.3]

2. Secondary Outcome: Response Rate (RR)
Description: Response Rate (RR) is defined as any patient whom has a documented complete response (CR) or partial response (PR) per RECIST version 1.1 criteria. Results will be reported by number of participants for each response type: CR or PR.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Complete Response | 0
  Partial Response | 0

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Median PFS will be calculated in months from date of first dose of protocol therapy to date of documented disease progression or death from any cause, where progression is defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as at least a 20% increase in the sum of the SLD of target lesions, taking as reference the smallest sum of the SLD recorded since the treatment started and minimum 5 millimeter (mm) increase over the nadir, or the appearance of one or more new lesions for target lesions and/or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Kaplan-Meier methods will be used to summarize time-to-event outcomes.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 28
months | 3.7 [2.2 to 5.3]

4. Secondary Outcome: Median Overall Survival (OS)
Description: Median OS for all enrolled patients (intention-to-treat) will be calculated from date of first dose of protocol therapy until date of death, using chart review and/or follow up phone calls to determine date of death in patients after removal from study. The survival of patients still alive after 5 years of follow up post study discontinuation will be censored.
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 28
months | 8.8 [6.8 to 14.8]

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF will be measured from date of first dose of protocol therapy to date of study discontinuation for progression, death, or toxicity.
Time Frame: 24 months
Measure: Median (Full Range); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 28
months | 3.1 [0.7 to 15]

6. Secondary Outcome: Number of Patients With a Demonstrated Alpha-fetoprotein (AFP) Response
Description: In patients with baseline AFP >= 20 ng/mL, AFP response will be measured by the percent change from baseline value to the value at the time of best AFP response. The number of participants with ≥ 50% decline from baseline will be measured.
Time Frame: 24 months
Population: Only 21 patients had AFP response data available at time of best AFP response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 21
Participants | 10

7. Secondary Outcome: Number of Patients Whom Required a Dose Reduction
Description: The number of patients whom required a dose reduction due to toxicity as classified by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be reported
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
Participants | 13

8. Secondary Outcome: Number of Patients Whom Required a Treatment Delay
Description: The number of patients whom required a treatment delay due to toxicity as classified by the CTCAE version 4.0 will be reported
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
Participants | 14

9. Secondary Outcome: Number of Participants Whom Discontinued Treatment Due to Intolerable Toxicity
Description: The number of participants whom discontinued treatment due to toxicity as classified by the CTCAE version 4.0 will be reported
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
Participants | 6

ADVERSE EVENTS:
Time Frame: Up to 60 months
Description: Only patients actively treated with a combination of Temsirolimus and Sorafenib were evaluated for safety.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 27/28
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 20/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=28)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=28)
Hypophosphatemia (Metabolism and nutrition disorders) | 17 (50)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Platelet count decreased (Investigations) | 10 (22)
Weight loss (Investigations) | 7 (11)
Blood bilirubin increased (Investigations) | 3 (5)
Cholesterol high (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (10)
Diarrhea (Gastrointestinal disorders) | 8 (11)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (4)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 7 (8)
Edema limbs (General disorders) | 6 (7)
Chills (General disorders) | 3 (3)
Infusion related reaction (General disorders) | 3 (5)
Fever (General disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (14)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 3 (10)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT01687673/Prot_SAP_000.pdf